CLINICAL TRIAL: NCT00630695
Title: Evaluation of the Efficacity of Lanreotide LP 90 mg to Minimized the Lymphorrhea Post Axillary Lymphadenectomy in Breast Cancer
Brief Title: Prevention of Lymphorrhea by Lanreotide in Axillary Dissection for Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Collaborators: Ipsen (Industry)
Responsible Party: CHU de Limoges, CHU de Limoges
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2007-003576-19
Record Dates: First submitted 2008-02-27; First posted 2008-03-07 (Estimated); Last update posted 2012-01-16 (Estimated); Status verified 2012-01

CONDITIONS: Lymphocele
Keywords: Axillary lymphocele breast cancer
MeSH Terms: conditions — Lymphocele

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Lanreotide LP 90
  Interventions: Drug: Lanreotide LP 90
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo lanreotide

INTERVENTIONS:
Drug: Lanreotide LP 90 — Lanreotide LP 90
  Arms: 1
Drug: Placebo lanreotide — Placebo
  Arms: 2

SUMMARY:
Injection the day before surgery of 90 mg of Lanreotide LP sub-cutaneously or placebo. Evaluation of the lymphorrhea in the 2 arms of the study

DETAILED DESCRIPTION:
Patients will be recruited among patient refered to our department for a breast cancer and needing an axillary dissection. Enrolled patients will have an injection of Lanreotide or placebo the day before surgery when they arrive in their room. The quantity of lymph in axillary drain will by daily noted until day 4. The patient will be evaluated at D15, D30 and M6 for pain, lymphocele and adverse events.

Data will be compared in the 2 groups.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (> 18 years),
* Patient undergoing an axillary lymphadenectomy for breast cancer
* Patient giving her agreement after being informed

Exclusion Criteria:

* Patients that don't understand the trial
* Type 2 diabetic patients
* Cyclosporine treatment
* Biliary lithiasis
* Pregnancy or breast feeding
* Allergic reaction to Lanréotide or same class treatments
* Patient included in another trial within the last 30 days

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2008-03; Primary Completion 2011-06 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Quantity of lymph collected by the drain | D4 post operativly

SECONDARY OUTCOMES:
Prevention of lymphocele | D15, D30 and M6

CONTACTS AND LOCATIONS:
Overall Officials: Yves Aubard, MD, PhD, Study Chair — University Hospital, Limoges
Locations (1):
- Hôpital Mère Enfant- CHU de Limoges, Limoges, France